CLINICAL TRIAL: NCT03922854
Title: Determining the Predictive Utility of Short-term Variation (STV) of Fetal Heart Rate (FHR) for Fetal Acidaemia, and the Feasibility of Using This for Decision Making in High-risk Women During Labour
Brief Title: Monitoring of Babies' Heart Rates During Labour Using Mobile Monitors
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH19362
Record Dates: First submitted 2018-08-14; First posted 2019-04-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Fetal Acidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mobile Monitor Group: Participants are recruited to this study if they have been monitored during their labour with a monica AN 24 monitor
  Interventions: Other: Non-interventional data collection only

INTERVENTIONS:
Other: Non-interventional data collection only — There is no clinical intervention. This study is just capturing data from devices used part of routine clinical care. The results of this data collection will be analysed to inform study results.

SUMMARY:
The study has been designed as a prospective, non-randomised, single centre study to determine the predictive utility of Short Term Variation (STV) of the Fetal Heart Rate (FHR)from the intrapartum FHR data collected using the portable fetal ECG monitor (Monica AN24) in women requiring continuous monitoring during labour due to antenatal or intrapartum risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Singleton term pregnant labouring women during established labour (cervix >3cm dilated, regular uterine contractions >3:10 minutes)
* Written informed consent
* At least 18 years of age

Exclusion Criteria:

* Preterm labouring women
* Multiple pregnancy
* Involved in another study using a device or medicinal product

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female pregnant and being given monicar in 204 monitor
Study Population: Pregnant population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Sample Size | Recruitment period January 2018-April 2019
  This is a feasibility study with a primary objective to establish design of a large multi-centre study. Outcome measure is percentage number of participants to have a umbilical blood cord gas PH level below 7.20. This will inform the statistical sample for the larger study.
Recruitment Rate | Recruitment period January 2018-April 2019
  This is a feasibility study with a primary objective to establish design of a large multi-centre study. Outcome measure is how many participants recruited per month this will inform how many centre's will be required to deliver statistical sample size for larger study.
Data Capture | Recruitment period January 2018-April 2019
  This is a feasibility study with a primary objective to establish design of a large multi-centre study. Outcome measure is number of completed data sets. A complete data set equals more than one hour of recorded data from mobile fetal heart rate monitor and arterial umbilical cord blood gas level taken. This will inform estimated sample size for larger study.

CONTACTS AND LOCATIONS:
Overall Officials: Habiba Kapaya, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Jessop Wing Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No